CLINICAL TRIAL: NCT05310968
Title: Study on Tirofiban With Aspirin in the Treatment of Acute Penetrating Artery Territory Infarction (STRATEGY)
Brief Title: Study on Tirofiban With Aspirin in the Treatment of Acute Penetrating Artery Territory Infarction
Acronym: STRATEGY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: GrandPharma (China) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2021-089-08
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Branch Atheromatous Disease
Keywords: branch atheromatous disease; perforating artery territorial infarction; tirofiban; aspirin; randomized controlled trial; multicenter study; double blind study; placebo-controlled
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): This group will receive tirofiban and aspirin. Day 1: Tirofiban injected intravenously for 24 hours and aspirin of 100-300 mg. Tirofiban will be injected at 0.4 ug/kg/ min for the first 30 minutes and 0.1 ug/kg/min for the next 24 hours.
  Day 2-90: Aspirin 100mg per day.
  Interventions: Drug: Tirofiban hydrochloride sodium chloride injection; Drug: Aspirin
- Tirofiban placebo group (Placebo Comparator): This group will receive tirofiban placebo and aspirin. Day 1: Tirofiban placebo injected intravenously for 24 hours and aspirin of 100-300 mg. The placebo will be injected at the same rate with Tirofiban group.
  Day 2-90: Aspirin 100mg per day.
  Interventions: Drug: Tirofiban hydrochloride sodium chloride injection placebo; Drug: Aspirin

INTERVENTIONS:
Drug: Tirofiban hydrochloride sodium chloride injection — Day 1: Tirofiban will be given by bolus injection at 0.4ug/kg/min for the first 30 minutes, followed by a continuous infusion at 0.1ug/kg/min for the next 24 hours.
  Arms: Tirofiban group
Drug: Tirofiban hydrochloride sodium chloride injection placebo — Day 1: Tirofiban placebo will be injected at the same rate with experimental group.
  Arms: Tirofiban placebo group
Drug: Aspirin — Day 1: Aspirin 100-300mg per day Day 2-90: Aspirin 100mg per day

SUMMARY:
Perforating artery territorial infarction (PAI) refers to a single ischemic lesion in a single perforating arterial territory and branch atheromatous disease (BAD) is an important type. BAD related stroke accounts for 10%-15% ischemic cerebral infarction and is closely related to early neurological deterioration (END). Among patients with single ischemic lesion in other study, dual antiplatelet (clopidogrel plus aspirin) did not significantly reduce the risk of recurrent stroke. The primary purpose of this study is to assess the efficacy and safety of tirofiban combined with aspirin versus placebo combined with aspirin in reducing the risk of stroke and END in patients with BAD.

DETAILED DESCRIPTION:
Branch atheromatous disease (BAD) was characterized by cerebral infarction within penetrating artery territories. It arises from atherosclerotic stenosis or occlusion at the origin or proximal segment of these arteries, with three principal pathological manifestations. BAD is the typical etiology of the isolated infarction in penetrating artery territories. There is still no consensus on the classification, and both the TOAST and the CISS (Chinese ischemic stroke subclassification) have the limitations.

Currently, there are no evidence-supported, guideline-based on how to prevent the END of BAD. Combining the pathology of atherosclerosis, we hypothesize that short-term use of tirofiban with aspirin for intensive antiplatelet therapy may confer benefits.

The primary purpose of this study is to assess the efficacy and safety of tirofiban combined with aspirin versus placebo combined with aspirin in reducing END and stroke at 90 days in patients with BAD.

This is a prospective, randomized, multicenter, double-blind clinical trial. In China, 970 patients with the following criteria will be enrolled: single acute infarction of penetrating artery territory (maximum diameter <30 mm on DWI of MRI) within 48 hours, which involves two or more transverse layers, or whose maximum diameter ≥15 mm, , or connected to the ventral surface of the median pons without crossing the midline on DWI image, no severe stenosis (defined as <70%) of parent artery.

Patients will be randomly assigned into 2 groups:

1. Tirofiban + Aspirin (Day 1-90)
2. Placebo + Aspirin (Day 1-90) Interviews will be made on baseline, 24 hours after randomization, day 7 after randomization, discharge day, and day 90 after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Male or female;
3. Within 48 hours of onset;
4. Clinical symptoms and signs suggest acute single infarction of penetrating artery territory (no cortical involvement, no multifocal involvement, NIHSS ≤10 and consciousness-1a ≤1);
5. DWI suggests single infarction (diameter < 30mm) of penetrating artery territory which involves at least 2 axial layers, or its maximum diameter ≥15mm, or it is connected to the ventral surface of the pons, closing to but not crossing the midline, and located in one side;
6. No severe stenosis (defined as <70%) of parent artery;
7. The patient or his / her legal representative is able and willing to sign the informed consent.

Exclusion Criteria:

1. History of intracranial hemorrhage
2. History of intracranial tumors, cerebral arteriovenous malformation, or aneurysm;
3. Emergency endovascular intervention or intravenous thrombolysis before randomization;
4. Dual antiplatelet therapy currently or within 14 days of randomization (excluding use of aspirin and clopidogrel after onset without loading dose of clopidogrel);
5. Use of other antiplatelet drugs (ticagrelor, cilostazol, etc.), anticoagulant drugs, snake venom, defibrase, lumbrukinase or other defibrase treatments after onset;
6. Expected long-term use of non-investigational antiplatelet drugs or non-steroidal anti-inflammatory drugs;
7. With severe stenosis (> 70%) of parent artery giving off responsible penetrating artery;
8. Definite indications for anticoagulation (suspicion of cardioembolism, e.g. atrial fibrillation, known heart valve prosthesis, atrial myxoma, endocarditis, etc.) or indications for dual antiplatelet therapy (e.g. recent coronary or cerebral artery stent implantation);
9. Severe hepatic or renal insufficiency before randomization (severe hepatic insufficiency refers to ALT or AST > 3 times the upper limit of normal; severe renal insufficiency refers to creatinine clearance rate (CCr) < 30ml/min);
10. Hemorrhagic tendency (including but not limited to)：PLT<100×10^9/L; heparin treatment within 48h; APTT ≥ 35s; current use of warfarin, INR > 1.7; current use of novel oral anticoagulants; current use of direct thrombin or factor Xa inhibitor;
11. Resistant hypertension which could not be controlled by medicine (SBP > 180mmHg or DBP > 110mmHg);
12. History of obvious head trauma within three months of randomization;
13. History of intracranial or intramedullary surgery within three months of randomization;
14. History of major surgery or severe physical trauma within one month of randomization;
15. Severe neurological defects (mRS ≥ 2) before the onset;
16. Acute pericarditis;
17. Hemorrhagic retinopathy;
18. Childbearing-age women who do not take effective methods of contraception without negative records of pregnancy tests;
19. Known to be allergic to tirofiban;
20. Other surgical or interventional therapy planned within 3 months requiring experimental drugs discontinuation;
21. Life expectancy < 6 months due to any terminal illness;
22. Patients who are undergoing experimental drugs or instruments;
23. Other conditions which suggest participants are unsuitable for this study, e.g. mental diseases, cognitive or mood disturbance,and could not comply with research procedures or with MRI contraindications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
new stroke or END(early neurological deterioration） | 90 days after randomization
  1. Symptoms and signs of acute neurological deficits caused by sudden focal or whole brain, spinal cord, or retinal vascular damage, which are related to cerebral circulatory disorders, including hemorrhagic and ischemic stroke.
  2. NIHSS score increasing by ≥ 2 points, or the score increasing by≥1 in either the motor or consciousness level within 7 days after randomization and intracranial hemorrhage is excepted by CT or MRI. Exacerbations not attributable to stroke are also excluded such as cardiac failure, liver and renal failure, etc.

SECONDARY OUTCOMES:
new stroke or END | 24 hours and 7 days after randomization
  1)Symptoms and signs of acute neurological deficits caused by sudden focal or whole brain, spinal cord, or retinal vascular damage, which are related to cerebral circulatory disorders, including hemorrhagic and ischemic stroke. 2)NIHSS score increasing by ≥ 2 points, or the score increasing by≥1 in either the motor or consciousness level within 7 days after randomization and intracranial hemorrhage is excepted by CT or MRI. Exacerbations not attributable to stroke are also excluded such as cardiac failure, liver and renal failure, etc.
Composite vascular events | 90 days after randomization
  Symptomatic stroke, myocardial infarction and vascular death.
Disability or death | 90 days after randomization
  The modified Rankin Scale (mRS) is 2-6 points.
Improvement of neurological function | 24 hours, 7 days, and 90 days after randomization
  decrease of NIHSS score by ≥4 points or NIHSS score of 0-1 point
EQ-5D-5L Scale | 90 days after randomization
  It describes the state of health.

OTHER OUTCOMES:
Moderate or severe bleeding events | 90 days after randomization
  Number of participants with Moderate or severe bleeding events
Symptomatic and non-symptomatic intracranial hemorrhage | 90 days after randomization
  According to Heidelberg Bleeding Classification.
Vascular death | 90 days after randomization
  Stroke, myocardial infarction, peripheral arterial ischemia, other vascular-related deaths and sudden death and unexplained death.
Overall mortality | 90 days after randomization
  The ratio of total deaths from all causes to the research subjects
Number of participants with dverse event/serious adverse event | 90 days after randomization
  PLT≤100×10^9/L; hypersensitivity; renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD，MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (37):
- China (37):
  - The First Hospital of Fangshan District Beijing, Beijing, Beijing Municipality
  - School of Medicine, Xiamen University, Zhangzhou, Fujian
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hejian People's Hospital, Hejian, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - The People's Hospital of Qinghe County, Xingtai, Hebei
  - Mengzhou People's Hospital, Henan, Henan
  - Xiuwu People's Hospital, Jiaozuo, Henan
  - Jiyuan Hospital of Traditional Chinese Medicine, Jiyuan, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Tanghe County People's Hospital, Nanyang, Henan
  - The First People's Hospital of Nanyang, Nanyang, Henan
  - Suixian Hospital of Traditional Chinese Medicine, Shangqiu, Henan
  - The People's Hospital of Biyang County, Zhumadian, Henan
  - Shaodong People's Hospital, Shaoyang, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The First Affiliate Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Affiliated Nantong Hospital of Shanghai University (The Sixth People's Hospital of Nantong), Nantong, Jiangsu
  - The People's Hospital of Suxitong Science & Technology Inductrial Park, Nantong, Jiangsu
  - The Affiliated Shuyang Hospital of Xuzhou Medical University, Suqian, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Benxi Central Hospital, Benxi, Liaoning
  - The First People's Hospital of Xianyang, Xianyang, Shaanxi
  - Ningjin People's Hospital, Dezhou, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Guanxian People's Hospital, Liaocheng, Shandong
  - Liaocheng Central Hospital, Liaocheng, Shandong
  - The People's Hospital of Gaotang County, Liaocheng, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - The Third People's Hospital of Liaocheng, Liaocheng, Shandong
  - The People's Hospital of Linqing, Linqing, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weihai Wendeng District People's Hospital, Weihai, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Jincheng People's Hospital, Jincheng, Shanxi
  - Wanrong County People's Hospital, Yuncheng, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu H, Howatt DA, Balakrishnan A, Graham MJ, Mullick AE, Daugherty A. Hypercholesterolemia Induced by a PCSK9 Gain-of-Function Mutation Augments Angiotensin II-Induced Abdominal Aortic Aneurysms in C57BL/6 Mice-Brief Report. Arterioscler Thromb Vasc Biol. 2016 Sep;36(9):1753-7. doi: 10.1161/ATVBAHA.116.307613. Epub 2016 Jul 28. PMID 27470509
- [Background] Seitz RJ, Meisel S, Moll M, Wittsack HJ, Junghans U, Siebler M. The effect of combined thrombolysis with rtPA and tirofiban on ischemic brain lesions. Neurology. 2004 Jun 8;62(11):2110-2. doi: 10.1212/01.wnl.0000129480.17345.4a. PMID 15184627
- [Background] Berberich A, Schneider C, Reiff T, Gumbinger C, Ringleb PA. Dual Antiplatelet Therapy Improves Functional Outcome in Patients With Progressive Lacunar Strokes. Stroke. 2019 Apr;50(4):1007-1009. doi: 10.1161/STROKEAHA.118.023789. PMID 30841818
- [Background] Coull AJ, Lovett JK, Rothwell PM; Oxford Vascular Study. Population based study of early risk of stroke after transient ischaemic attack or minor stroke: implications for public education and organisation of services. BMJ. 2004 Feb 7;328(7435):326. doi: 10.1136/bmj.37991.635266.44. Epub 2004 Jan 26. PMID 14744823
- [Background] Jeong HG, Kim BJ, Yang MH, Han MK, Bae HJ. Neuroimaging markers for early neurologic deterioration in single small subcortical infarction. Stroke. 2015 Mar;46(3):687-91. doi: 10.1161/STROKEAHA.114.007466. Epub 2015 Feb 12. PMID 25677600
- [Background] Cohen JE, Rabinstein A, Gomori JM, Leker RR. Capsular warning syndrome and crescendo lacunar strokes after atherosclerotic stenosis of the recurrent artery of Heubner. J Clin Neurosci. 2012 Dec;19(12):1730-3. doi: 10.1016/j.jocn.2012.04.010. Epub 2012 Sep 19. PMID 22999563
- [Background] Del Bene A, Palumbo V, Lamassa M, Saia V, Piccardi B, Inzitari D. Progressive lacunar stroke: review of mechanisms, prognostic features, and putative treatments. Int J Stroke. 2012 Jun;7(4):321-9. doi: 10.1111/j.1747-4949.2012.00789.x. Epub 2012 Mar 30. PMID 22463492
- [Background] Sudlow CL, Warlow CP. Comparable studies of the incidence of stroke and its pathological types: results from an international collaboration. International Stroke Incidence Collaboration. Stroke. 1997 Mar;28(3):491-9. doi: 10.1161/01.str.28.3.491. PMID 9056601
- [Background] Caplan LR. Lacunar infarction and small vessel disease: pathology and pathophysiology. J Stroke. 2015 Jan;17(1):2-6. doi: 10.5853/jos.2015.17.1.2. Epub 2015 Jan 30. PMID 25692102
- [Background] Bang OY. Intracranial atherosclerosis: current understanding and perspectives. J Stroke. 2014 Jan;16(1):27-35. doi: 10.5853/jos.2014.16.1.27. Epub 2014 Jan 31. PMID 24741562
- [Background] Kim BJ, Kim JS. Ischemic stroke subtype classification: an asian viewpoint. J Stroke. 2014 Jan;16(1):8-17. doi: 10.5853/jos.2014.16.1.8. Epub 2014 Jan 31. PMID 24741560
- [Background] Kim JS, Yoon Y. Single subcortical infarction associated with parental arterial disease: important yet neglected sub-type of atherothrombotic stroke. Int J Stroke. 2013 Apr;8(3):197-203. doi: 10.1111/j.1747-4949.2012.00816.x. Epub 2012 May 9. PMID 22568537
- [Background] Fisher CM. Capsular infarcts: the underlying vascular lesions. Arch Neurol. 1979 Feb;36(2):65-73. doi: 10.1001/archneur.1979.00500380035003. PMID 420625
- [Background] Caplan LR. Intracranial branch atheromatous disease: a neglected, understudied, and underused concept. Neurology. 1989 Sep;39(9):1246-50. doi: 10.1212/wnl.39.9.1246. No abstract available. PMID 2671793
- [Derived] Liao X, Feng S, Wang Y, Pan Y, Chen W, Qu H, Zhao X, Liu L, Wang Y, Wang Y. Tirofiban combined with Aspirin in the Treatment of Acute Penetrating Artery Territory Infarction (STRATEGY): protocol for a multicentre, randomised controlled trial. Stroke Vasc Neurol. 2024 Feb 27;9(1):75-81. doi: 10.1136/svn-2022-002284. PMID 37220998